CLINICAL TRIAL: NCT01810185
Title: Low Dose Naltrexone in Symptomatic Inflammatory Bowel Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Low patient enrollment
Sponsor: Santa Barbara Cottage Hospital (Other)
Responsible Party: Principal Investigator, Erick Jordan Imbertson, M.D., Santa Barbara Cottage Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LDN in IBD; SBCH- LDN in IBD (Other: Santa Barbara Cottage Hospital)
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: Inflammatory Bowel Disease; Crohn's disease; Ulcerative colitis; Naltrexone; Low Dose Naltrexone; Inflammatory Bowel Disease Questionnaire
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose naltrexone (Experimental): Subjects in this arm will recieve low dose naltrexone (4.5 mg) daily for 12 weeks.
  Interventions: Drug: Low dose naltrexone
- Placebo (Placebo Comparator): Subjects in this arm will recieve a placebo daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose naltrexone — 4.5 mg daily for 12 weeeks
  Other Names: Naltrexone
  Arms: Low dose naltrexone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The investigators will be looking at the efficacy of the use of once daily use of low dose naltrexone (4.5mg) in subjects with symptomatic inflammatory bowel disease.

DETAILED DESCRIPTION:
The investigators will compare the use of daily low dose naltrexone (LDN) (4.5 mg) compared with placebo in subjects that have symptomatic inflammatory bowel disease (IBD). Our subjects will be those with diagnosed with IBD and are symptomatic, defined by an inflammatory bowel disease questionnaire (IBDQ) score < 170. The subjects will be randomly assigned either placebo or LDN. They will take the IBDQ prior to starting the trial, 6 weeks, 12 weeks and 6 months after starting the medication. Participants have to remain on their current IBD regimen throughout the trial and cannot make any changes within 4 weeks of starting the trial. The investigators will have a safety phone call at 6 weeks and a follow up letter at 12 weeks after starting the trial. The participants will be given a card to keep with them with a phone number and email address if any adverse effects arise.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic Crohn's disease or ulcerative colitis (defined as a response to the Inflammatory Bowel Disease Questionnaire less than 170)
* Confirmed Crohn's disease or ulcerative colitis through radiographic, endoscopic and/or histologic criteria
* On a stable dose of medication for IBD (i.e. no change in medication within 4 weeks of study enrollment)
* Age 18 or older

Exclusion Criteria:

* Patients on opioids or immodium within 7 days of starting the investigational therapy
* Women who are breastfeeding, pregnant, or plan on becoming pregnant within the next year
* Patients on Lomotil or opioid analgesics
* Patients already on low dose naltrexone
* Women of child bearing age not willing to use contraception or abstinence
* A history of the following diseases or procedures:

  * Acute hepatitis
  * Liver failure
  * Ileoanal anastomosis
  * Short bowel syndrome
  * Abnormal liver enzymes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
An increase in the subjects inflammatory bowel disease questionnaire score | 6 weeks, 12 weeks, and 6 months
  Participants will fill-out a questionnaire called the IBDQ at enrollment, 6 weeks, 12 weeks, and 6 months after enrollment. The IBDQ is a validated instrument often used in routine care and studies of patients with IBD (Appendix E). The IBDQ measures the activity of IBD and quality of life. It includes 32 questions placed into 4 domains: bowel, social, emotional and systemic. Each question is ranked from 1-7, 1 being the poorest quality of life and 7 being the best quality of life8. A score of >170 means that a patient is clinically in remission and an increase in score between 16 and 32 are considered a meaningful improvement in symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Erick J Imbertson, M.D., Principal Investigator — Santa Barabara Cottage Hospital
Locations (1):
- Santa Barbara Cottage Hospital, Santa Barbara, California, United States

REFERENCES:
- [Result] Smith JP, Stock H, Bingaman S, Mauger D, Rogosnitzky M, Zagon IS. Low-dose naltrexone therapy improves active Crohn's disease. Am J Gastroenterol. 2007 Apr;102(4):820-8. doi: 10.1111/j.1572-0241.2007.01045.x. Epub 2007 Jan 11. PMID 17222320
- [Result] Smith JP, Field D, Bingaman SI, Evans R, Mauger DT. Safety and tolerability of low-dose naltrexone therapy in children with moderate to severe Crohn's disease: a pilot study. J Clin Gastroenterol. 2013 Apr;47(4):339-45. doi: 10.1097/MCG.0b013e3182702f2b. PMID 23188075
- [Result] Low-dose naltrexone: tricking the body to heal itself. Exp Biol Med (Maywood). 2011 Sep;236(9):vii-viii. doi: 10.1258/ebm.2011.011f08. No abstract available. PMID 21991594
- [Derived] Segal D, Macdonald JK, Chande N. Low dose naltrexone for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2014 Feb 21;(2):CD010410. doi: 10.1002/14651858.CD010410.pub2. PMID 24558033